CLINICAL TRIAL: NCT07005037
Title: Improving Recovery in Older ICU Survivors: Evaluation of Swallowing Dysfunction and Aspiration Risk
Brief Title: Swallowing Impairments in ICU Survivors and Community-Dwelling Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cara Donohue, Ph.D. CCC-SLP, Assistant Professor, Director of Medical Speech-Language Pathology, Vanderbilt University Medical Center
Other Study IDs: 250839
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Dysphagia; Healthy Aging; Post Intensive Care Syndrome; Caregiver Burden
MeSH Terms: conditions — Deglutition Disorders; postintensive care syndrome; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy community dwelling adults: Healthy community dwelling adults who meet the inclusion criteria for the study will be enrolled.
- ICU survivors and their care partners: Critically ill adults and their care partners who meet inclusion criteria for the study will be enrolled.

SUMMARY:
Post-intensive care syndrome (PICS), which consists of physical, cognitive, and psychosocial problems, is a pervasive complication for older intensive care unit (ICU) survivors and contributes to detrimental health outcomes and significant reductions in quality of life. Yet, little is known about the relationship between PICS, swallowing difficulties (dysphagia), and other ICU-related negative outcomes such as frailty and Alzheimer's Disease and Related Dementias (ADRD). The primary purpose of this research study is to determine the prevalence and severity of dysphagia, risk factors for dysphagia development, recovery patterns of dysphagia over time, and the impact of dysphagia on health outcomes, quality of life, and care partner burden in adult ICU survivors with PICS.

DETAILED DESCRIPTION:
This study will involve one in-person research visit for community dwelling adults and two research visits for critically ill adults (one in the ICU, one 3-months post-hospital discharge) that will last approximately 1 hour and will consist of a screening, cough testing, swallow function testing, assessments of hand grip and tongue strength, and completion of questionnaires. Caregivers of ICU survivors will complete questionnaires at the 3-month follow up visit.

ELIGIBILITY:
Inclusion criteria community-dwelling adults:

1. adult ≥18 years old
2. no prior history of neurological diseases or respiratory diseases
3. no prior history of head and neck surgery/head and neck cancer/radiation to head and neck region
4. no prior history of dysphagia.

Exclusion criteria community-dwelling adults:

1. <18 years old
2. neurological disease or respiratory disease diagnosis
3. history of head and neck cancer/surgery to the head and neck region
4. history of dysphagia.

Inclusion criteria critically-ill adults:

1. adult ≥ 18 years old
2. ICU patients requiring monitoring or treatment for respiratory failure and/or shock (e.g., hypovolemic, septic, and/or cardiogenic)
3. cognitive capacity and willingness to provide informed consent
4. medically stable for testing (e.g., can sit upright, respiratory status is stable [Sp02 > 90%, off mechanical ventilation or CPAP/BiPAP for > 30 minutes, respiratory rate < 30 bpm], and Richmond Agitation-Sedation Scale score is 0 (awake and alert).

Exclusion criteria critically ill adults:

1. neurological disease diagnosis
2. history of head and neck cancer/surgery to the head and neck region
3. history of dysphagia prior to ICU admission.

Inclusion criteria caregivers:

1. caregiver of critically ill adult who meets inclusion criteria for study
2. willing to complete questionnaire.

Exclusion criteria caregivers:

1. not a caregiver of critically ill adult
2. unwilling to complete questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll 100 community dwelling adults who meet inclusion criteria, 180 critically ill adults who meet inclusion criteria, and 180 caregivers of critically ill adults who meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Swallowing safety and efficiency | During baseline visit at time of enrollment for community dwelling adults. During baseline visit at time of enrollment and 3 months post-hospital discharge for critically ill adults.
  The validated Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) scale will be used to measure swallowing safety and efficiency.

SECONDARY OUTCOMES:
Voluntary cough peak expiratory flow | During baseline visit at time of enrollment for community dwelling adults. During baseline visit at time of enrollment and 3 months post-hospital discharge for critically ill adults.
  A measure of cough strength
Grip strength | During baseline visit at time of enrollment for community dwelling adults. During baseline visit at time of enrollment and 3 months post-hospital discharge for critically ill adults.
  Grip strength be used to quantify clinical frailty using a digital hand dynamometer.
Tongue strength | During baseline visit at time of enrollment for community dwelling adults. During baseline visit at time of enrollment and 3 months post-hospital discharge for critically ill adults.
  Tongue strength will be assessed using the Iowa Oral Pressure Instrument (IOPI).
Swallowing and Eating Related Fatigue Questionnaire (SERF) | During baseline visit at time of enrollment for community dwelling adults. During baseline visit at time of enrollment and 3 months post-hospital discharge for critically ill adults.
  Scores on the SERF range 0-48 with higher scores indicating greater impairment.
Eating Assessment Tool 10 (EAT-10) | During baseline visit at time of enrollment for community dwelling adults. During baseline visit at time of enrollment and 3 months post-hospital discharge for critically ill adults.
  The EAT-10 contains 10 questions (score range: 0-40), higher scores indicate greater impairment.
3 oz water swallow test | During baseline visit at time of enrollment for community dwelling adults. During baseline visit at time of enrollment and 3 months post-hospital discharge for critically ill adults.
  Participants will be given a cup of three ounces of water and instructed to drink the water continuously. Fail criteria includes interrupted drinking and/or coughing/throat clearing during or immediately following the drinking task.
Reflex cough | During baseline visit at time of enrollment for community dwelling adults. During baseline visit at time of enrollment and 3 months post-hospital discharge for critically ill adults.
  Participants will undergo reflex cough testing.
Screening for Oral Frailty Tool (SOFT) | During baseline visit at time of enrollment for community dwelling adults. During baseline visit at time of enrollment and 3 months post-hospital discharge for critically ill adults.
  Oral frailty will be assessed as present/absent using the Screening for Oral Frailty Tool.
Swallowing Related Quality of Life Questionnaire (SWAL-QOL) | During baseline visit at time of enrollment for community dwelling adults. 3 months post-hospital discharge for critically ill adults.
  Scores on the SWAL-QOL range from 0-100 with lower scores indicating greater impairment.
Caregiver Analysis of Reported Experiences with Swallowing Disorders (CARES) Questionnaire | 3 months post-hospital discharge for care partners of critically ill adults.
  Scores on the CARES range from 0-26 with higher scores indicating greater caregiver burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No